CLINICAL TRIAL: NCT03137225
Title: Noninvasive NAVA Versus NIPPV in Low Birthweight Premature Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources available to complete the study
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM20005575
Record Dates: First submitted 2017-04-17; First posted 2017-05-02 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Noninvasive Ventilation; Low Birth Weight
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Intervention Model Description: Randomization - the order of modes will be assigned based on a random number table using a 5 block design to match the DSMB reporting needs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nasal Intermittent Positive Pressure Ventilation (NIPPV) Mode (Experimental): After a one hour stabilization period, during which small adjustments to the noninvasive settings can be made to clinically optimize the settings, the study will begin. A Nellcor pulse oximeter probe will be placed on an extremity to provide a continuous non-invasive downloadable measure of saturation (blood oxygen level) and heart rate. Data from the ventilator will be downloaded in real-time to a laptop.
  These data will be recorded for 4 hours continuously. After that, the ventilator will be switched to the other mode (NIPPV to NAVA), at the same PEEP (positive end-expiratory pressure) and respiratory rate. One hour will be allowed to adjust the ventilator settings. Data will then be collected for 4 hours on the second ventilation mode (NAVA)
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Nasal Intermittent Positive Pressure Ventilation
- Neurally Adjusted Ventilatory Assist (NAVA) Mode (Experimental): After a one hour stabilization period, during which small adjustments to the noninvasive settings can be made to clinically optimize the settings, the study will begin. A Nellcor pulse oximeter probe will be placed on an extremity to provide a continuous non-invasive downloadable measure of saturation (blood oxygen level) and heart rate. Data from the ventilator will be downloaded in real-time to a laptop.
  These data will be recorded for 4 hours continuously. After that, the ventilator will be switched to the other mode (NAVA to NIPPV), at the same PEEP and respiratory rate. One hour will be allowed to adjust the ventilator settings. Data will then be collected for 4 hours on the second ventilation mode (NIPPV)
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Nasal Intermittent Positive Pressure Ventilation

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist — Neurally Adjusted Ventilatory Assist delivered via RAM cannula .
  Other Names: NAVA
Device: Nasal Intermittent Positive Pressure Ventilation — Nasal Intermittent Positive Pressure Ventilation delivered via RAM cannula
  Other Names: NIPPV

SUMMARY:
The investigator hypothesizes that in very low birth weight infants who require respiratory support via noninvasive ventilation, that synchronizing the ventilator breath with the baby's breath using neurally adjusted ventilatory assist (NAVA) will reduce the number and/or severity of apnea/bradycardia/desaturation episodes compared to nasal intermittent positive pressure ventilation (NIPPV).

DETAILED DESCRIPTION:
Very low birthweight (VLBW) premature infants in the NICU (Neonatal Intensive Care Unit) frequently require respiratory support for prolonged periods of time. Invasive mechanical ventilation (which requires intubating the baby with a tube to provide breaths) can lead to ventilator induced lung injury. Because of this, noninvasive respiratory support has become increasingly popular, as this form of ventilation has been shown to reduce the incidence of permanent lung injury.

There are several methods to provide non-invasive support. The gentlest is continual flow of air and oxygen via nasal cannula. However, premature infants often develop apnea, either because the signals from their immature brain are not yet sufficient or because the muscles in the back of their throat do not get enough nerve signals to maintain sufficient opening. As a result, babies on nasal cannula often develop clinical apnea/bradycardia/desaturations. Before putting these babies back on invasive ventilation, clinicians often try to provide the baby with machine breaths while still on non-invasive ventilation.

This method is called nasal intermittent positive pressure ventilation and studies have demonstrated that this method reduces the need for re-intubation in VLBW infants (1) and reduces the rate of apneic events.

A newer method of non-invasive breathing support that has been FDA approved and used in VLBW infants, synchronizes the machine generated breath with the patient's own breath. Neurally adjusted ventilatory assist (NAVA) does this by replacing the standard nasogastric tube with a nasogastric tube that has sensors which detect the baby's natural diaphragm activity, which signal the ventilator to breath in synchronization with the baby. Studies have shown that the efficacy of nasal ventilation is significantly enhanced when the machine breath is synchronized with the patient breath (2). Synchronization also reduces diaphragmatic dysfunction (3). It can improve gas delivery, reduce work of breathing, and make patients demonstrably more comfortable (4).

Neurally Adjusted Ventilatory Assist (NAVA) is a mode of partial support. NAVA can be used both in intubated patients (invasive NAVA) as well as in extubated patients who require noninvasive positive pressure ventilation (noninvasive NAVA) (5). Invasive NAVA has been shown to deliver equivalent ventilation while requiring lower peak inspiratory pressure, as well as reduced respiratory muscle load, compared to conventional pressure support ventilation.

Currently, the choice of using NIPPV or NAVA is at the clinician's discretion. Both are regularly and frequently used in the VCU (Virginia Commonwealth University) Health System's NICU. There are no studies that have examined whether NAVA triggered synchronized ventilation is more effective than nonsynchronized NIPPV. In addition, there is limited data on the synchronicity and mechanics of non-invasive NAVA in VLBW infants. Information comparing clinical and lung mechanical outcomes between NIPPV and NIV (Nasal noninvasive ventilation) NAVA would significantly benefit VLBW care providers and, consequently, their patients in getting the best evidenced based therapy.

ELIGIBILITY:
Inclusion Criteria:

* < 1501 grams (VLBW (very low birth weight) infant)
* Patient must be receiving daily caffeine therapy for apnea
* On non-invasive ventilation, either NIPPV or non-invasive NAVA

Exclusion Criteria:

* No concerns for acute sepsis (i.e., blood cultures, if drawn, have been negative for 48 hours, and no active signs/symptoms of sepsis).
* No history of meningitis or seizures
* No signs of increased intracranial pressure, including bulging fontaneIle, presence of ventricular shunt device, or ventriculomegaly by most recent ultrasound.
* Presence of Grade III or IV intraventricular hemorrhage
* No cyanotic heart defects or clinically significant congenital heart disease. Will allow PDA (patent ductus arteriosus), PFO (patent foramen ovale), and mild to moderate ASD (atrial septal defect)/VSD (ventricular septal defect) as determined by pediatric cardiology.
* Non -English speaking legal representatives (parents)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry J Rozycki, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang S, Zhao J, Shen J, Hu Z, Shi Y. Nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure in neonates: a systematic review and meta-analysis. Indian Pediatr. 2013 Apr;50(4):371-6. doi: 10.1007/s13312-013-0122-0. Epub 2012 Oct 5. PMID 23255684
- [Result] Gizzi C, Montecchia F, Panetta V, Castellano C, Mariani C, Campelli M, Papoff P, Moretti C, Agostino R. Is synchronised NIPPV more effective than NIPPV and NCPAP in treating apnoea of prematurity (AOP)? A randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2015 Jan;100(1):F17-23. doi: 10.1136/archdischild-2013-305892. Epub 2014 Oct 15. PMID 25318667
- [Result] Petrof BJ, Jaber S, Matecki S. Ventilator-induced diaphragmatic dysfunction. Curr Opin Crit Care. 2010 Feb;16(1):19-25. doi: 10.1097/MCC.0b013e328334b166. PMID 19935062
- [Result] Stein H, Firestone K. Application of neurally adjusted ventilatory assist in neonates. Semin Fetal Neonatal Med. 2014 Feb;19(1):60-9. doi: 10.1016/j.siny.2013.09.005. Epub 2013 Nov 13. PMID 24238745
- [Result] Moerer O, Beck J, Brander L, Costa R, Quintel M, Slutsky AS, Brunet F, Sinderby C. Subject-ventilator synchrony during neural versus pneumatically triggered non-invasive helmet ventilation. Intensive Care Med. 2008 Sep;34(9):1615-23. doi: 10.1007/s00134-008-1163-z. Epub 2008 May 30. PMID 18512045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Groups:
- NIPPV Then NAVA Mode: After a one hour stabilization period, during which small adjustments to the noninvasive settings can be made to clinically optimize the settings, the study will begin. A Nellcor pulse oximeter probe will be placed on an extremity to provide a continuous non-invasive downloadable measure of saturation (blood oxygen level) and heart rate. Data from the ventilator will be downloaded in real-time to a laptop.
  The ventilator will be set Nasal Intermittent Positive Pressure Ventilation (NIPPV) mode.
  These data will be recorded for 4 hours continuously. After that, the ventilator will be switched to Neurally Adjusted Ventilatory Assist (NAVA) mode, at the same PEEP (positive end-expiratory pressure) and respiratory rate.
  One hour will be allowed to adjust the ventilator settings. Data will then be collected for 4 hours on the second ventilation mode (NAVA)
- NAVA Then NIPPV Mode: After a one hour stabilization period, during which small adjustments to the noninvasive settings can be made to clinically optimize the settings, the study will begin. A Nellcor pulse oximeter probe will be placed on an extremity to provide a continuous non-invasive downloadable measure of saturation (blood oxygen level) and heart rate. Data from the ventilator will be downloaded in real-time to a laptop.
  The ventilator will be set to Neurally Adjusted Ventilatory Assist (NAVA) mode. These data will be recorded for 4 hours continuously. After that, the ventilator will be switched to Nasal Intermittent Positive Pressure Ventilation (NIPPV) mode , at the same PEEP (positive end-expiratory pressure) and respiratory rate.
  One hour will be allowed to adjust the ventilator settings. Data will then be collected for 4 hours on the second ventilation mode.
Period: First 4 Hour Measurement Period
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Second 4 Hour Measurement Period
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 subject enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: participants] — Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Unexpected Events
Description: The number of isolated apneas, bradycardias and desaturations and the number of combined events will be compared by mode of ventilation.
Time Frame: 8 hours - from placement on first study ventilation mode to the end of the second study ventilation mode.
Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Synchronicity
Description: Synchronicity from the ventilator at the time of an event. This will be analyzed to determine whether asynchronicity is related to increased number of events during the study.
Time Frame: 8 hours - from placement on first study ventilation mode to the end of the second study ventilation mode.
Population: as for outcome 1
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Asynchronicity Counts
Description: Overall asynchronicity counts will be determined by ventilator data that can be uploaded and analyzed with software supplied by the manufacturer.
Time Frame: During each four hour treatment segment
Population: as for outcome 1
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Average Pressures
Description: Average mean airway pressure and peak inspiratory pressures required in each mode of ventilation.
Time Frame: 8 hours - from placement on first study ventilation mode to the end of the second study ventilation mode.
Population: as for outcome 1
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 hours
Arm/Group | NIPPV Then NAVA Mode | NAVA Then NIPPV Mode
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT03137225/Prot_SAP_000.pdf